CLINICAL TRIAL: NCT04068792
Title: A Two-Part Study With a Birth Cohort (Observational Stage) for Early Diagnosis of Respiratory Syncytial Virus (RSV), Followed by an Optional Phase 2a, Randomized, Double-blind, Placebo-controlled Study (Interventional Stage) to Evaluate the Antiviral Activity, Clinical Outcomes, Safety, Tolerability, and Pharmacokinetics of JNJ-53718678 in Infants With Acute Respiratory Tract Infection Due to RSV
Brief Title: A Two-Part Infant Study for Early Diagnosis of Respiratory Syncytial Virus (RSV) and Evaluation of JNJ-53718678 in RSV Acute Respiratory Tract Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108647; 2019-001509-25 (EudraCT Number); 53718678RSV2006 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Results first posted 2022-06-08 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Respiratory Syncytial Viruses
MeSH Terms: interventions — JNJ-53718678

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Part 1-Observational Phase (Other): Participants will not receive any intervention in the observation phase. All infants will be closely monitored for early signs and symptoms of Respiratory Syncytial Virus (RSV) disease using a mobile RSV application on the parent/caregiver's mobile phone, upon an alert, the RSV will be tested, if RSV negative participants (RSV [-] diagnosed at site) will return to the pre-diagnostic phase and RSV positive participants (RSV [+] diagnosed at site) can be enrolled in the interventional stage of the study after obtaining informed consent for the interventional stage at that time. RSV (+) participants whose parent(s)/caregiver(s) do not consent for enrollment in the interventional stage and participants who are screening failures in the interventional stage will enter the post-diagnostic phase of the observational stage (hospitalized or outpatients).
  Interventions: Other: RSV Mobile Application
- Part 2-Interventional Phase (Experimental): Participants will be randomized to receive either JNJ-53718678 (for Age Group 1 (greater than or equal to [>=] 28 days and less than [<] 3 months): 2.5 milligram per kilogram [mg/kg]; for Age Group 2 (>=3 and <6 months): 3 mg/kg and for Age Group 3 (>=6 months): 4.5 mg/kg) or placebo (Age Group 1, 2 and 3) twice daily for 7 days.
  Interventions: Drug: Placebo; Drug: JNJ-53718678 2.5 mg/kg; Drug: JNJ-53718678 3 mg/kg; Drug: JNJ-53718678 4.5 mg/kg

INTERVENTIONS:
Other: RSV Mobile Application — Participants will not receive any intervention in observational phase of this study. Participant's respiratory symptoms will be captured by RSV mobile application installed in participant's caregiver/parent mobile phone.
  Arms: Part 1-Observational Phase
Drug: Placebo — Participants in each Age Group (1,2,3) will receive matching placebo (volume placebo to match the calculated volume of the JNJ-53718678 dose) orally twice daily for 7 days.
  Arms: Part 2-Interventional Phase
Drug: JNJ-53718678 2.5 mg/kg — JNJ-53718678 will be administered to Age Group 1 twice daily for 7 days.
  Arms: Part 2-Interventional Phase
Drug: JNJ-53718678 3 mg/kg — JNJ-53718678 will be administered to Age Group 2 twice daily for 7 days.
  Arms: Part 2-Interventional Phase
Drug: JNJ-53718678 4.5 mg/kg — JNJ-53718678 will be administered to Age Group 3 twice daily for 7 days.
  Arms: Part 2-Interventional Phase

SUMMARY:
The purpose of this two-part designed study is to assess in the setting of a planned early interception of pediatric RSV disease, early viral and disease kinetics (observational stage) and the antiviral effects of an Respiratory Syncytial Virus (RSV) fusion inhibitor, JNJ-53718678 (interventional stage). In the observational stage the infant is closely monitored for early symptoms by the parent(s)/caregiver(s) and thus may be brought in for diagnosis earlier than in the typical setting.

ELIGIBILITY:
Inclusion Criteria:

Part 1: Observational Stage

* The infant is less than or equal to (<=) 4 months of age at enrollment and asymptomatic for acute respiratory illness (ARI)-like symptoms requiring medical intervention at the time of consent to participate in the study
* At least 1 parent/caregiver must be able to use the respiratory syncytial virus (RSV) mobile application (App) at home via his/her own Android/iOS electronic device (compatible with RSV mobile App)
* The participant must have been assessed per local public health practice and considered not to have Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection

Part 2: Interventional Stage

* The infant is 28 days and if prematurely born infant (that is [i.e.], less than [<] 37 weeks and 0 days of gestation at birth) is at least 3 months postnatal age
* The participant has been diagnosed with RSV infection using a rapid molecular-based diagnostic assay
* The participant weighs more than 2.4 kilogram (kg)
* The participant has an acute respiratory illness as evaluated by the investigator
* Except for the RSV-related illness, the participant must be medically stable in case of allowed co-morbid conditions
* The participant must have been assessed per local public health practice and considered not to have SARS-CoV-2 infection during this respiratory infection

Exclusion Criteria:

Part 1: Observational Stage

* The participant has any physical abnormality which limits the ability to collect regular nasal specimens
* The participant is receiving chronic home oxygen therapy at enrollment (applicable to both parts)

Part 2: Interventional Stage

* The participant is <3 months postnatal age at screening and was born prematurely (i.e., <37 weeks and 0 days of gestation) or if the participant weights <2.4 kg
* The participant has a QT interval with Fridericia's correction (QTcF) greater than (>) 450 milliseconds per the machine read (mean of triplicate) parameter result confirmed by repeat triplicate Electrocardiogram (ECG) recording during screening
* The participant is considered by the investigator to be immunocompromised, whether due to underlying medical condition or medical therapy
* The participant has had any of: a) Confirmed SARS-CoV-2 infection (test positive) during the four weeks prior to randomization, or b) Close contact with a person with Coronavirus Disease 2019 (COVID-19) (test confirmed or suspected SARS-CoV-2 infection) within 14 days prior to randomization

Ages: 28 Days to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (10):
- Instituto de Maternidad y Ginecología Nuestra Senora de las Mercedes, San Miguel de Tucumán, Argentina
- UZ Antwerpen, Edegem, Belgium
- Panama (3):
  - Cevaxin 24 de diciembre, Panama City
  - Cevaxin Avenida Mexico, Panama City
  - Cevaxin La Chorrera, Republica de Panama
- Taiwan (4):
  - Hsinchu MacKay Memorial Hospital, Hsinchu
  - National Taiwan University Hospital, Taipei
  - Department of Pediatrics, MacKay Memorial Hospital, Taipei
  - Chang Gung Memorial Hospital- Linkou, Taoyuan District
- St George's University Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinicaltrials/ transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: As per original dosing, participants were randomized to receive JNJ-53718678 matching placebo (for Age Group 1 [greater than or equal to {>=} 28 days and less than {<} 3 months], for Age Group 2 [>=3 and <6 months], and for Age Group 3 [>=6 months]) orally once daily (qd) for 7 days. After Protocol amendment 2, participants were randomized to receive JNJ-53718678 matching placebo (for Age Groups 1, 2, and 3) orally twice daily (bid) for 7 days.
- JNJ-53718678: As per original dosing, participants were randomized to receive JNJ-53718678 (for Age Group 1 [>= 28 days and < 3 months]: 5 milligrams/kilogram [mg/kg]; for Age Group 2 [>=3 and <6 months]: 6 mg/kg and for Age Group 3 [>=6 months]: 9 mg/kg) orally qd for 7 days. After Protocol amendment 2, participants were randomized to receive JNJ-53718678 (for Age Group 1: 2.5 mg/kg; for Age Group 2: 3 mg/kg and for Age Group 3: 4.5 mg/kg) orally bid for 7 days
Period: Overall Study
Arm/Group | Placebo | JNJ-53718678
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | JNJ-53718678 | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: months] | 4.10 (1.962) | 3.18 (1.343) | 3.64 (1.707)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 8 | 7 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 10 | 8 | 18
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 0 | 1 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Panama | 11 | 10 | 21
  Taiwan, Province Of China | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Respiratory Syncytial Virus (RSV) Viral Load-time Curve From Immediately Prior to First Dose of JNJ-53718678 Through Day 5 (AUC [Day 1-5])
Description: RSV viral load AUC was determined from immediately prior to first dose of JNJ-53718678 through Day 5. The RSV viral load was measured by quantitative reverse transcription polymerase chain reaction (qRT-PCR) assay in mid-turbinate nasal swab specimens.
Time Frame: Baseline (Day 1) up to Day 5
Population: Intent-To-Treat-infected (ITT-i) analysis set included all randomized participants who received at least one dose of study drug and who had a centrally confirmed RSV viral load of greater than or equal to (>=) 1 log10 copies per milliliter (mL) above the lower limit of quantification (LLOQ) of the RSV RT-qPCR assay at baseline. Analyses on the ITT-i set were performed as randomized.
Measure: Mean (90% Confidence Interval); unit: log10 copies*day per milliliter
Arm/Group | Placebo | JNJ-53718678
Number analyzed (Participants) | 11 | 10
log10 copies*day per milliliter | 26.13 (23.701) [23.701 to 28.555] | 25.10 (22.497) [22.497 to 27.707]
Statistical Analysis 1: Comparison: Placebo vs JNJ-53718678; Test type: Other; Mean Difference (Final Values) = -1.03, 90% CI 2-sided [-4.467 to 2.416]

2. Secondary Outcome: RSV Viral Load Over Time
Description: RSV viral load actual values over time was measured by qRT-PCR in the nasal swab specimens collected at the clinic visits and at home.
Time Frame: Baseline, Days 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, and 21
Population: ITT-i analysis set included all randomized participants who received at least one dose of study drug and who had a centrally confirmed RSV viral load of >= 1 log10 copies per mL above the LLOQ of the RSV RT-qPCR assay at baseline. Analyses on the ITT-i set were performed as randomized. Here 'n' (number analyzed) included all participants who were analyzed at specified timepoints.
Measure: Mean (Standard Deviation); unit: log10 copies per milliliter
Arm/Group | Placebo | JNJ-53718678
Number analyzed (Participants) | 11 | 10
log10 copies per milliliter
  Baseline | 7.744 (1.1991) | 7.477 (1.4111)
  Day 2: number analyzed (Participants) | 10 | 7
  Day 2 | 7.748 (1.2387) | 6.613 (3.2426)
  Day 3: number analyzed (Participants) | 11 | 9
  Day 3 | 6.415 (2.3924) | 6.277 (2.8027)
  Day 4: number analyzed (Participants) | 9 | 8
  Day 4 | 5.600 (2.2868) | 5.683 (3.2009)
  Day 5: number analyzed (Participants) | 11 | 6
  Day 5 | 6.105 (1.3664) | 5.287 (2.0195)
  Day 6: number analyzed (Participants) | 10 | 6
  Day 6 | 4.335 (2.3774) | 4.023 (2.8076)
  Day 7: number analyzed (Participants) | 8 | 6
  Day 7 | 4.953 (1.0500) | 3.624 (2.4153)
  Day 8: number analyzed (Participants) | 9 | 8
  Day 8 | 4.020 (0.9431) | 2.924 (2.1366)
  Day 9: number analyzed (Participants) | 5 | 4
  Day 9 | 3.145 (1.8643) | 2.666 (2.1545)
  Day 10: number analyzed (Participants) | 4 | 4
  Day 10 | 2.657 (1.9192) | 3.035 (2.2622)
  Day 11: number analyzed (Participants) | 5 | 3
  Day 11 | 2.598 (1.6655) | 3.059 (2.6895)
  Day 12: number analyzed (Participants) | 3 | 3
  Day 12 | 0.967 (1.6743) | 3.417 (3.4191)
  Day 14: number analyzed (Participants) | 9 | 8
  Day 14 | 2.352 (2.3700) | 2.020 (2.4599)
  Day 21: number analyzed (Participants) | 11 | 9
  Day 21 | 1.837 (1.9135) | 0.883 (1.3426)

3. Secondary Outcome: Change From Baseline in RSV Viral Load Over Time
Description: Change from baseline in RSV viral load over time was measured by qRT-PCR in the nasal swab specimens collected at the clinic visits and at home.
Time Frame: Baseline, Days 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, and 21
Population: ITT-i analysis set included all randomized participants who received at least one dose of study drug and who had a centrally confirmed RSV viral load of >= 1 log10 copies per mL above the LLOQ of the RSV RT-qPCR assay at baseline. Analyses on the ITT-i set were performed as randomized. Here, 'n' (number analyzed) included all participants who were analyzed at specified timepoints.
Measure: Mean (Standard Deviation); unit: log10 copies per milliliter
Arm/Group | Placebo | JNJ-53718678
Number analyzed (Participants) | 11 | 10
log10 copies per milliliter
  Day 2: number analyzed (Participants) | 10 | 7
  Day 2 | 0.022 (0.9247) | -0.797 (1.8465)
  Day 3: number analyzed (Participants) | 11 | 9
  Day 3 | -1.329 (2.3903) | -1.293 (1.6220)
  Day 4: number analyzed (Participants) | 9 | 8
  Day 4 | -2.002 (2.7624) | -1.857 (1.9805)
  Day 5: number analyzed (Participants) | 11 | 6
  Day 5 | -1.638 (1.4728) | -2.222 (1.4063)
  Day 6: number analyzed (Participants) | 10 | 6
  Day 6 | -3.391 (2.8796) | -3.153 (1.5444)
  Day 7: number analyzed (Participants) | 8 | 6
  Day 7 | -2.667 (1.8529) | -3.552 (1.1919)
  Day 8: number analyzed (Participants) | 9 | 8
  Day 8 | -3.630 (1.5622) | -4.634 (1.6078)
  Day 9: number analyzed (Participants) | 5 | 4
  Day 9 | -5.046 (1.8708) | -5.564 (2.2160)
  Day 10: number analyzed (Participants) | 4 | 4
  Day 10 | -5.782 (2.3406) | -5.195 (2.3057)
  Day 11: number analyzed (Participants) | 5 | 3
  Day 11 | -5.580 (1.8008) | -5.263 (2.7523)
  Day 12: number analyzed (Participants) | 3 | 3
  Day 12 | -7.225 (0.9469) | -4.905 (3.4450)
  Day 14: number analyzed (Participants) | 9 | 8
  Day 14 | -5.439 (2.0248) | -5.588 (2.7565)
  Day 21: number analyzed (Participants) | 11 | 9
  Day 21 | -5.907 (1.6829) | -6.514 (1.5001)

4. Secondary Outcome: RSV Viral Load Area Under the Curve (AUC) From Immediately Prior to First Dose of Study Drug (Baseline) Through Days 3, 8, and 14
Description: RSV viral load AUC was determined by qRT-PCR assay in mid-turbinate nasal swab specimens.
Time Frame: Baseline through Days 3, 8, and 14
Population: ITT-i analysis set included all randomized participants who received at least one dose of study drug and who had a centrally confirmed RSV viral load of >=1 log10 copies per mL above the LLOQ of the RSV RT-qPCR assay at baseline. Analyses on the ITT-i set was performed as randomized. Here 'n' (number analyzed) included all participants who were analyzed at specified timepoints. At Day 14, data was not collected due to low sample size.
Measure: Mean (90% Confidence Interval); unit: log10 copies*hour per milliliter (h/mL)
Arm/Group | Placebo | JNJ-53718678
Number analyzed (Participants) | 11 | 10
log10 copies*hour per milliliter (h/mL)
  Day 3 | 14.44 [12.841 to 16.042] | 13.70 [11.990 to 15.406]
  Day 8 | 39.20 [34.913 to 43.491] | 35.11 [31.342 to 38.880]
  Day 14: number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Time to Undetectable RSV Viral Load
Description: Time to undetectable RSV viral load is defined as the time in hours from initiation of study treatment until the first post-baseline time point at which the virus is confirmed undetectable. A confirmed undetectable sample is defined as the first of at least two consecutive samples that are undetectable. The last obtained sample for a participant, if undetectable, is considered confirmed.
Time Frame: Up to 21 days
Population: ITT-i analysis set included all randomized participants who received at least one dose of study drug and who had centrally confirmed RSV viral load of >=1 log10 copies per mL above the LLOQ of the RSV RT-qPCR assay at baseline. Analyses on the ITT-i set was performed as randomized.
Measure: Median (90% Confidence Interval); unit: hours
Arm/Group | Placebo | JNJ-53718678
Number analyzed (Participants) | 11 | 10
hours | 500.1 [239.90 to NA] — 'NA' refers that upper limit of confidence interval was not estimable due to low sample size, and censoring. | 391.4 [185.50 to 526.20]

6. Secondary Outcome: Percentage of Participants With Undetectable RSV Viral Load at Each Time Point Throughout the Study
Description: Percentage of participants with undetectable RSV viral load at each time point throughout the study were reported.
Time Frame: Baseline, Days 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 21
Population: ITT-i analysis set included all randomized participants who received at least one dose of study drug and who had a centrally confirmed RSV viral load of >=1 log10 copies per mL above the LLOQ of the RSV RT-qPCR assay at baseline. Analyses on the ITT-i set was performed as randomized. Here 'n' (number analyzed) included all participants who were analyzed at specified timepoints.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | JNJ-53718678
Number analyzed (Participants) | 11 | 10
percentage of participants
  Baseline | 0 | 0
  Day 2: number analyzed (Participants) | 10 | 7
  Day 2 | 0 | 14.3
  Day 3: number analyzed (Participants) | 11 | 9
  Day 3 | 9.1 | 11.1
  Day 4: number analyzed (Participants) | 9 | 8
  Day 4 | 11.1 | 12.5
  Day 5: number analyzed (Participants) | 11 | 6
  Day 5 | 0 | 0
  Day 6: number analyzed (Participants) | 10 | 6
  Day 6 | 20.0 | 16.7
  Day 7: number analyzed (Participants) | 8 | 6
  Day 7 | 0 | 16.7
  Day 8: number analyzed (Participants) | 9 | 8
  Day 8 | 0 | 25.0
  Day 9: number analyzed (Participants) | 5 | 4
  Day 9 | 20.0 | 25.0
  Day 10: number analyzed (Participants) | 4 | 4
  Day 10 | 25.0 | 25.0
  Day 11: number analyzed (Participants) | 5 | 3
  Day 11 | 20.0 | 33.3
  Day 12: number analyzed (Participants) | 3 | 3
  Day 12 | 66.7 | 33.3
  Day 14: number analyzed (Participants) | 9 | 8
  Day 14 | 33.3 | 50.0
  Day 21: number analyzed (Participants) | 11 | 9
  Day 21 | 45.5 | 66.7

7. Secondary Outcome: Severity of Signs and Symptoms of RSV Infection Assessed by Parent(s)/Caregiver(s) Pediatric RSV Electronic Severity and Outcome Rating System (PRESORS)
Description: The severity of signs and symptoms of RSV infection (breathing problems, retractions, tachypnea, breathing sounds, cough, tachycardia, nasal secretions, sleep disturbance, crying, illness behavior, feeding problems, and dehydration) were assessed by the PRESORS. PRESORS is a questionnaire by parent(s)/caregiver(s) recording presence and severity of signs and symptoms of RSV disease. PRESORS score consisted of 12-items, each score ranges from 0 to 3. A summary score was derived (mean of the item scores) which also ranges from 0 to 3. The higher the score, the worse the symptom.
Time Frame: Baseline, Days 3, 5, 8, 14, and 21
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Unit on scale
Arm/Group | Placebo | JNJ-53718678
Number analyzed (Participants) | 11 | 10
Unit on scale
  Baseline: number analyzed (Participants) | 10 | 8
  Baseline | 0.92 (0.345) | 0.56 (0.527)
  Day 3: number analyzed (Participants) | 11 | 8
  Day 3 | 0.98 (0.535) | 0.60 (0.610)
  Day 5: number analyzed (Participants) | 11 | 9
  Day 5 | 0.65 (0.456) | 0.37 (0.398)
  Day 8 | 0.61 (0.461) | 0.23 (0.285)
  Day 14 | 0.14 (0.323) | 0.08 (0.162)
  Day 21: number analyzed (Participants) | 10 | 10
  Day 21 | 0.15 (0.337) | 0.02 (0.053)

8. Secondary Outcome: Change From Baseline in Parent(s)/Caregiver(s) PRESORS Scores
Description: PRESORS is a questionnaire recording presence and severity of signs and symptoms of RSV disease. PRESORS score consisted of 12-items, each item score ranges from 0 to 3. A summary score was derived (mean of the item scores) which also ranges from 0 to 3. The higher the score, the worse the symptom.
Time Frame: Baseline, Day 3, 5, 8, 14, 21
Population: ITT-i analysis set included all randomized participants who received at least one dose of study drug and who had a centrally confirmed RSV viral load of >=1 log10 copies per mL above the LLOQ of the RSV RT-qPCR assay at baseline. Analyses on the ITT-i set were performed as randomized. Here 'N' (number of participants analyzed), included all participants who were evaluable for this outcome measure. Here 'n' (number analyzed) included all participants who were analyzed at specified timepoints.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Placebo | JNJ-53718678
Number analyzed (Participants) | 10 | 8
units on scale
  Day 3: number analyzed (Participants) | 10 | 7
  Day 3 | 0.01 (0.341) | -0.02 (0.249)
  Day 5 | -0.27 (0.309) | -0.26 (0.437)
  Day 8 | -0.42 (0.314) | -0.39 (0.508)
  Day 14 | -0.73 (0.396) | -0.54 (0.396)
  Day 21: number analyzed (Participants) | 9 | 8
  Day 21 | -0.70 (0.408) | -0.60 (0.390)

9. Secondary Outcome: Change From Baseline in Clinician PRESORS Score
Description: Change from baseline in clinician (for concepts: activity level, sleep disturbance, breathing problems, retractions, tachypnea, feeding problem, cough, nasal secretions, wheezing, dehydration) PRESORS scores was reported. PRESORS is a questionnaire recording presence and severity of signs and symptoms of RSV disease. PRESORS score consisted of 10-items, each item score ranges from 0 to 3. A summary score was derived (mean of the item scores) which also ranges from 0 to 3. The higher the score, the worse the symptom.
Time Frame: Baseline, Day 3, 5, 8, 14, 21
Population: ITT-i analysis set included all randomized participants who received at least one dose of study drug and who had centrally confirmed RSV viral load of >=1 log10 copies per mL above LLOQ of RSV RT-qPCR assay at baseline. Analyses on ITT-i set were performed as randomized. Here 'N' (number of participants analyzed), included all participants who were evaluable for this outcome measure; 'n' (number analyzed) included all participants who were analyzed at specified timepoints for specific category.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Placebo | JNJ-53718678
Number analyzed (Participants) | 9 | 7
units on scale
  Day 3: number analyzed (Participants) | 8 | 7
  Day 3 | 0.03 (0.287) | 0.01 (0.212)
  Day 5 | -0.32 (0.291) | -0.04 (0.162)
  Day 8 | -0.36 (0.167) | -0.16 (0.151)
  Day 14: number analyzed (Participants) | 9 | 6
  Day 14 | -0.42 (0.192) | -0.10 (0.192)
  Day 21 | -0.42 (0.192) | -0.24 (0.276)

10. Secondary Outcome: Time to Resolution of RSV Symptoms
Description: Time to resolution from first dose of study drug until the first time of resolution of all RSV Symptoms (breathing problems, retractions, tachypnea, breathing sounds, cough, tachycardia, nasal secretions, sleep disturbance, crying, illness behavior, feeding problems, and dehydration). Resolution occurs when all symptoms from the caregiver reported outcomes (ObsRO) are scored as none or mild (score of 0 or 1, respectively) for at least 24 hours.
Time Frame: Up to 21 days
Population: ITT-i analysis set included all randomized participants who received at least one dose of study drug and who had a centrally confirmed RSV viral load of >=1 log10 copies per mL above the LLOQ of the RSV RT-qPCR assay at baseline. Analyses on the ITT-i set were performed as randomized.
Measure: Median (90% Confidence Interval); unit: Hours
Arm/Group | Placebo | JNJ-53718678
Number analyzed (Participants) | 11 | 10
Hours | 194.00 [164.20 to 238.00] | 118.60 [17.00 to 238.00]

11. Secondary Outcome: Time to Improvement on Overall Health
Description: Time to improvement based on general questions on overall health was reported. Time from first dose of study drug until first time status of improvement of RSV symptoms reported as "very much improved" or "much improved" based on response to question 'Would you say the child's RSV symptoms have improved, are about the same or are worse than when the child entered the study'.
Time Frame: Up to 21 days
Population: ITT-i analysis set included all randomized participants who received at least one dose of study drug and who had a centrally confirmed RSV viral load of >=1 log10 copies per mL above the LLOQ of the RSV RT-qPCR assay at baseline. Analyses on the ITT-i set was performed as randomized.
Measure: Median (90% Confidence Interval); unit: Hours
Arm/Group | Placebo | JNJ-53718678
Number analyzed (Participants) | 11 | 10
Hours | 188.3 [183.60 to 238.00] | 199.7 [183.70 to 238.00]

12. Secondary Outcome: Percentage of Participants With Worsening or Improvement of RSV Disease
Description: Percentage of participants with worsening or improvement of RSV disease based on general questions on overall health was reported. Improvement is defined improvement of RSV symptoms reported as "very much improved" or "much improved" based on response to question 'Would you say the child's RSV symptoms have improved, are about the same or are worse than when the child entered the study'.
Time Frame: On Days 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21
Population: ITT-i analysis set included all randomized participants who received at least one dose of study drug and who had a centrally confirmed RSV viral load of >=1 log10 copies per mL above the LLOQ of the RSV RT-qPCR assay at baseline. Analyses on the ITT-i set were performed as randomized. Here 'n' (number analyzed) included all participants who were analyzed at specified timepoints.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | JNJ-53718678
Number analyzed (Participants) | 11 | 10
percentage of participants
  Day 2 : Very Much Improved: number analyzed (Participants) | 3 | 1
  Day 2 : Very Much Improved | 0 | 0
  Day 2: Very Much Worse: number analyzed (Participants) | 3 | 1
  Day 2: Very Much Worse | 0 | 0
  Day 3: Very Much Improved: number analyzed (Participants) | 3 | 1
  Day 3: Very Much Improved | 0 | 0
  Day 3: Very Much Worse: number analyzed (Participants) | 3 | 1
  Day 3: Very Much Worse | 0 | 0
  Day 4: Very Much Improved: number analyzed (Participants) | 3 | 1
  Day 4: Very Much Improved | 0 | 0
  Day 4: Very Much Worse: number analyzed (Participants) | 3 | 1
  Day 4: Very Much Worse | 0 | 0
  Day 5: Very Much Improved: number analyzed (Participants) | 3 | 1
  Day 5: Very Much Improved | 0 | 0
  Day 5: Very Much Worse: number analyzed (Participants) | 3 | 1
  Day 5: Very Much Worse | 0 | 0
  Day 6: Very Much Improved: number analyzed (Participants) | 3 | 1
  Day 6: Very Much Improved | 66.7 | 0
  Day 6: Very Much Worse: number analyzed (Participants) | 3 | 1
  Day 6: Very Much Worse | 0 | 0
  Day 7: Very Much Improved: number analyzed (Participants) | 3 | 1
  Day 7: Very Much Improved | 66.7 | 0
  Day 7: Very Much Worse: number analyzed (Participants) | 3 | 1
  Day 7: Very Much Worse | 0 | 0
  Day 8: Very Much Improved: number analyzed (Participants) | 3 | 2
  Day 8: Very Much Improved | 33.3 | 50.0
  Day 8: Very Much Worse: number analyzed (Participants) | 3 | 2
  Day 8: Very Much Worse | 0 | 0
  Day 9: Very Much Improved: number analyzed (Participants) | 10 | 7
  Day 9: Very Much Improved | 60 | 42.9
  Day 9: Very Much Worse: number analyzed (Participants) | 10 | 7
  Day 9: Very Much Worse | 0 | 0
  Day 10: Very Much Improved | 36.4 | 50.0
  Day 10 Very Much Worse | 0 | 0
  Day 11 Very Much Improved: number analyzed (Participants) | 11 | 8
  Day 11 Very Much Improved | 54.5 | 37.5
  Day 11: Very Much Worse: number analyzed (Participants) | 11 | 8
  Day 11: Very Much Worse | 0 | 0
  Day 12 Very Much Improved: number analyzed (Participants) | 11 | 8
  Day 12 Very Much Improved | 54.5 | 62.5
  Day 12: Very Much Worse: number analyzed (Participants) | 11 | 8
  Day 12: Very Much Worse | 0 | 0
  Day 13 Very Much Improved | 90.0 | 50.0
  Day 13: Very Much Worse | 0 | 0
  Day 14: Very Much Improved: number analyzed (Participants) | 11 | 9
  Day 14: Very Much Improved | 90.0 | 55.6
  Day 14: Very Much Worse: number analyzed (Participants) | 11 | 9
  Day 14: Very Much Worse | 0 | 0
  Day 15: Very Much Improved: number analyzed (Participants) | 11 | 7
  Day 15: Very Much Improved | 90.9 | 57.1
  Day 15: Very Much Worse: number analyzed (Participants) | 11 | 7
  Day 15: Very Much Worse | 0 | 0
  Day 16: Very Much Improved: number analyzed (Participants) | 9 | 10
  Day 16: Very Much Improved | 77.8 | 80.0
  Day 16: Very Much Worse: number analyzed (Participants) | 9 | 10
  Day 16: Very Much Worse | 0 | 0
  Day 17: Very Much Improved: number analyzed (Participants) | 8 | 9
  Day 17: Very Much Improved | 87.5 | 88.9
  Day 17: Very Much Worse: number analyzed (Participants) | 8 | 9
  Day 17: Very Much Worse | 0 | 0
  Day 18: Very Much Improved: number analyzed (Participants) | 9 | 10
  Day 18: Very Much Improved | 88.9 | 80.0
  Day 18: Very Much Worse: number analyzed (Participants) | 9 | 10
  Day 18: Very Much Worse | 0 | 0
  Day 19: Very Much Improved: number analyzed (Participants) | 10 | 8
  Day 19: Very Much Improved | 90.0 | 75.0
  Day 19: Very Much Worse: number analyzed (Participants) | 10 | 8
  Day 19: Very Much Worse | 0 | 0
  Day 20: Very Much Improved: number analyzed (Participants) | 9 | 10
  Day 20: Very Much Improved | 88.9 | 70.0
  Day 20: Very Much Worse: number analyzed (Participants) | 9 | 10
  Day 20: Very Much Worse | 0 | 0
  Day 21: Very Much Improved: number analyzed (Participants) | 9 | 9
  Day 21: Very Much Improved | 88.9 | 77.8
  Day 21: Very Much Worse: number analyzed (Participants) | 9 | 9
  Day 21: Very Much Worse | 0 | 0

13. Secondary Outcome: Time to Return to Pre-RSV Health as Rated by the Parent(s)/Caregiver(s)
Description: Time to return to pre-RSV health as rated by the parent(s)/caregiver(s) was evaluated. It is the time from first dose of study drug until the time to return to pre-RSV disease level.
Time Frame: Up to 21 days
Population: Data was not collected due to low number of participants. Hence, no results are reported.
Arm/Group | Placebo | JNJ-53718678
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Percentage of Participants Who Require (re)Hospitalization During Treatment and Follow-up
Description: Percentage of participants who require (re)hospitalization during treatment and follow-up were reported.
Time Frame: Up to Day 31
Population: The Safety set (SAF) included all participants who received at least 1 dose of study drug, and were analyzed as treated, regardless of the randomized treatment group assigned. Where 'analyzed as treated' is defined as: Placebo: if only placebo doses received, and JNJ-53718678: if at least one dose of the active study drug received.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | JNJ-53718678
Number analyzed (Participants) | 11 | 11
Percentage of participants | 0 | 0

15. Secondary Outcome: Percentage of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Time Frame: Up to Day 31
Population: The SAF included all participants who received at least 1 dose of study drug, and were analyzed as treated, regardless of the randomized treatment group assigned. Where 'analyzed as treated' is defined as: Placebo: if only placebo doses received, and JNJ-53718678: if at least one dose of the active study drug received.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | JNJ-53718678
Number analyzed (Participants) | 11 | 11
percentage of participants | 27.3 | 27.3

16. Secondary Outcome: Percentage of Participants With Abnormal Chemistry Laboratory Findings
Description: Percentage of participants with abnormal chemistry laboratory findings (alanine aminotransferase [ALT; Grade 1 and 4], aspartate aminotransferase [AST; Grade 1], and Hyperkalemia [Grade 1 and 2]) were reported based on Division of Microbiology and Infectious Diseases (DMID) toxicity grading scale. DMID toxicity grades ranges from 1 to 4. Grade 1 = mild: transient or mild discomfort (<48 hours); no medical intervention/therapy required. Grade 2 = moderate: mild to moderate limitation in activity - some assistance may be needed; no or minimal medical intervention/therapy required. Grade 3 = severe: marked limitation in activity, some assistance usually required; medical intervention/therapy required, hospitalizations possible. Grade 4 = life-threatening or death: Extreme limitation in activity, significant assistance required; significant medical intervention/therapy required, hospitalization or hospice care probable.
Time Frame: Up to Day 31
Population: The SAF included all participants who received at least 1 dose of study drug, and were analyzed as treated, regardless of the randomized treatment group assigned. Where 'analyzed as treated' is defined as: Placebo: if only placebo doses received, and JNJ-53718678: if at least one dose of the active study drug received. Here 'n' (number analyzed) included all participants who were analyzed at specified categories.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | JNJ-53718678
Number analyzed (Participants) | 11 | 11
percentage of participants
  ALT Increase - Grade 1 | 9.1 | 0
  ALT Increase - Grade 4 | 9.1 | 0
  AST- Grade 1 | 9.1 | 18.2
  Hyperkalemia - Grade 1: number analyzed (Participants) | 10 | 11
  Hyperkalemia - Grade 1 | 30.0 | 0
  Hyperkalemia - Grade 2: number analyzed (Participants) | 10 | 11
  Hyperkalemia - Grade 2 | 10.0 | 0

17. Secondary Outcome: Percentage of Participants With Abnormal Urinalysis Laboratory Findings
Description: Percentage of participants with abnormal urinalysis (Hematuria- Grade 1) laboratory finding was reported based on DMID toxicity grading scale. DMID toxicity grades ranges from 1 to 4. Grade 1 = mild: transient or mild discomfort (<48 hours); no medical intervention/therapy required. Grade 2 = moderate: mild to moderate limitation in activity - some assistance may be needed; no or minimal medical intervention/therapy required. Grade 3 = severe: marked limitation in activity, some assistance usually required; medical intervention/therapy required, hospitalizations possible. Grade 4 = life-threatening or death: Extreme limitation in activity, significant assistance required; significant medical intervention/therapy required, hospitalization or hospice care probable.
Time Frame: Up to Day 31
Population: The SAF included all participants who received at least 1 dose of study drug, and were analyzed as treated, regardless of the randomized treatment group assigned. Where 'analyzed as treated' is defined as: Placebo: if only placebo doses received, and JNJ-53718678: if at least one dose of the active study drug received. Here 'N' (number of participants analyzed), included all participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | JNJ-53718678
Number analyzed (Participants) | 4 | 4
percentage of participants | 0 | 25.0

18. Secondary Outcome: Percentage of Participants With Abnormal Electrocardiograms (ECGs) Findings
Description: Percentage of participants with abnormal ECGs findings were reported. Parameters for abnormal ECG findings were QT interval corrected for heart rate (QTc) according to Bazett's formula (QTcB) Interval ([450 milliseconds {ms}, 480 ms], [480 ms, 500 ms], and [more than 500 ms]), QTc according to Fridericia's formula (QTcF) Interval ([450 ms, 480 ms], [480 ms, 500 ms], and [more than 500 ms]), change from baseline for QTcB Interval ([30; 60] ms, and greater than [>] 60 ms), and for QTcF Interval ([30; 60] ms, and >60 ms).
Time Frame: Up to Day 31
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | JNJ-53718678
Number analyzed (Participants) | 10 | 11
percentage of participants
  QTcB Interval (450 ms, 480 ms) | 20.0 | 9.1
  QTcB Interval (480 ms, 500 ms) | 0 | 0
  QTcB Interval (More than 500 ms) | 0 | 0
  QTcF Interval (450 ms, 480 ms) | 0 | 0
  QTcF Interval (480 ms, 500 ms) | 0 | 0
  QTcF Interval (More than 500 ms) | 0 | 0
  QTcB Interval (30; 60) ms | 0 | 9.1
  QTcB Interval (>60 ms) | 0 | 0
  QTcF Interval (30; 60) ms | 0 | 9.1
  QTcF Interval (>60 ms) | 0 | 0

19. Secondary Outcome: Percentage of Participants With Vital Sign Abnormalities
Description: Percentage of participants with vital signs (systolic blood pressure [SBP], diastolic blood pressure [DBP], pulse rate, respiratory rate, body temperature and peripheral capillary oxygen saturation [SpO2]) abnormalities (abnormally low [ABL] and abnormally high [ABH]) were reported.
Time Frame: Up to Day 31
Population: The SAF included all participants who received at least 1 dose of study drug, and were analyzed as treated, regardless of the randomized treatment group assigned. Where 'analyzed as treated' is defined as: Placebo: if only placebo doses received, and JNJ-53718678: if at least one dose of the active study drug received. Here 'n' (number analyzed) included all participants who were analyzed for specified categories.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | JNJ-53718678
Number analyzed (Participants) | 11 | 11
percentage of participants
  SBP- ABL: number analyzed (Participants) | 11 | 10
  SBP- ABL | 9.1 | 0
  SBP- ABH: number analyzed (Participants) | 11 | 10
  SBP- ABH | 0 | 0
  DBP- ABL: number analyzed (Participants) | 11 | 10
  DBP- ABL | 9.1 | 0
  DBP- ABH: number analyzed (Participants) | 11 | 10
  DBP- ABH | 0 | 0
  Pulse rate- ABL | 0 | 0
  Pulse rate- ABH | 9.1 | 18.2
  Respiratory Rate-ABL | 9.1 | 0
  Respiratory Rate-ABH | 0 | 0
  Temperature-ABL | 0 | 0
  Temperature-ABH | 27.3 | 45.5
  Oxygen Saturation- ABL: number analyzed (Participants) | 10 | 6
  Oxygen Saturation- ABL | 0 | 0
  Oxygen Saturation- ABH: number analyzed (Participants) | 10 | 6
  Oxygen Saturation- ABH | 0 | 0

20. Secondary Outcome: Plasma Concentrations of JNJ-53718678
Description: No data was collected for pharmacokinetic (PK) analysis due to small sample size. Hence, no results are reported.
Time Frame: Day 1 and Day 3
Population: No data was collected for PK analysis due to small sample size. Hence, no results are reported.
Arm/Group | Placebo | JNJ-53718678
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Day 31
Description: The safety analysis set (SAF) included all participants who were analyzed as treated, regardless of the randomized treatment group assigned for interventional stage. For interventional stage, 'analyzed as treated' is defined as; Placebo: if only placebo doses received, and JNJ-53718678: if at least one dose of the active study drug received.
Arm/Group | Placebo | JNJ-53718678
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 1/11 | 1/11
Other Adverse Events (participants affected / at risk) | 3/11 | 2/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=11) | JNJ-53718678 (N=11)
Respiratory Syncytial Virus Bronchiolitis (Infections and infestations) | 1 | 1
Tracheobronchitis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=11) | JNJ-53718678 (N=11)
Tachycardia (Cardiac disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 1
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis Diaper (Skin and subcutaneous tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The required number of participants in the interventional phase was not reached, and hence, limiting the interpretability of the data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2020-07-13): https://cdn.clinicaltrials.gov/large-docs/92/NCT04068792/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-02): https://cdn.clinicaltrials.gov/large-docs/92/NCT04068792/SAP_001.pdf